CLINICAL TRIAL: NCT00791739
Title: Open Label Trial Concerning the Effectiveness of Trazodone in the Treatment of Fibromyalgia (Phase I) and Its Augmentation With Pregabalin in Trazodone Partial Responders (Phase II)
Brief Title: Trazodone and Its Augmentation With Pregabalin in the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Elena Pita Calandre, Professor of Pharmacology, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TZD-PGB-2008
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; trazodone; pregabalin; Fibromyalgia Impact Questionnaire (FIQ); Pittsburgh Sleep Quality Inventory (PSQI); Brief Pain Inventory (BPI)
MeSH Terms: conditions — Fibromyalgia | interventions — Trazodone; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one arm study (Experimental)
  Interventions: Drug: trazodone, pregabalin

INTERVENTIONS:
Drug: trazodone, pregabalin — * phase I (from baseline to week 12): trazodone, in a starting dose of 50 mg at bedtime subsequently adjusted according to drug's efficacy and tolerability
  * phase II (from week 12 to week 24): addition of pregabalin in a starting dose of 75 mg/day subsequently adjusted according to drug's efficacy and tolerability
  Other Names: Deprax; Lyrica

SUMMARY:
The study has a double purpose: a first phase intends to assess the effectiveness and tolerability of trazodone, an antidepressant with sedative and sleep-promoting properties, in the treatment of fibromyalgia; a second phase intends to evaluate if the addition of pregabalin to patients who have shown a partial response to trazodone additionally improves fibromyalgia symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed of fibromyalgia according to the American College of Rheumatology criteria
* written, informed consent
* able to understand and comply with the requirements of the study

Exclusion Criteria:

* pregnancy or breastfeeding
* unwillingness to discontinue other prescribed medications before entering in the study
* patients who had previously received trazodone without improvement or who did not tolerate the drug
* patients who had previously received pregabalin without improvement or who did not tolerate the drug (only for the phase II of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Mean decrease, from baseline to endpoint, in the Fibromyalgia Impact Questionnaire | Baseline, 6, 12, 18 and 24 weeks

SECONDARY OUTCOMES:
Change from baseline to endpoint in the scores of the Pittsburgh Sleep Quality Inventory, the Brief Pain Inventory, the Beck Depression Inventory, and the Hospital Anxiety and Depression Scale | Baseline, 6, 12, 18, and 24 weeks
Discontinuation rates due to treatment-related adverse events, proportion of patients experiencing any adverse event, proportion of patients experiencing serious adverse events | baseline, 6, 12, 18, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elena P Calandre, MD, Principal Investigator — Universidad de Granada
Locations (1):
- Instituto de Neurociencias, Granada, Granada, Spain

REFERENCES:
- [Result] Morillas-Arques P, Rodriguez-Lopez CM, Molina-Barea R, Rico-Villademoros F, Calandre EP. Trazodone for the treatment of fibromyalgia: an open-label, 12-week study. BMC Musculoskelet Disord. 2010 Sep 10;11:204. doi: 10.1186/1471-2474-11-204. PMID 20831796
- [Derived] Calandre EP, Morillas-Arques P, Molina-Barea R, Rodriguez-Lopez CM, Rico-Villademoros F. Trazodone plus pregabalin combination in the treatment of fibromyalgia: a two-phase, 24-week, open-label uncontrolled study. BMC Musculoskelet Disord. 2011 May 16;12:95. doi: 10.1186/1471-2474-12-95. PMID 21575194
- See also: Web page of the Institute of Neuroscience of the University of Granada — http://www.ugr.es/~ineurociencias/ie/inicio.php